CLINICAL TRIAL: NCT02315742
Title: Healing Hearts and Mending Minds in Older Persons Living With HIV
Brief Title: Hearts and Minds in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rebecca Gary, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076644
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: HIV
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Let's Move Program (Experimental): Patients will take part in a 12-week exercise program.
  Interventions: Behavioral: Let's Move Program

INTERVENTIONS:
Behavioral: Let's Move Program — Patients will walk 5 times per week for 12 weeks for a minimum of 30 minutes while using a heart rate monitor. After the first two weeks of walking, patients will attend four consecutive group meetings which a research team member will look at walking logs and download data from heart rate monitor to focus on progress. Patient will receive weekly phone calls to monitor progress and to change walking duration or intensity level.
  Other Names: Exercise program

SUMMARY:
The purpose of this study is to see if walking is effective for improving memory, concentration thinking abilities, physical function and quality of life of adults 50 years of age and older living with HIV.

DETAILED DESCRIPTION:
By 2015 more than half of persons living with HIV (PLWH) in the U.S. will be older than 50 years of age. Two factors contribute to the "graying" of the HIV epidemic. The overwhelming success of antiretroviral therapy (ART) has improved life expectancy and dramatically changed the trajectory of HIV; it is now a complex chronic condition, often associated with multiple comorbidities such as cardiovascular disease (CVD) and cognitive impairment (CI). Second, increasing numbers of middle-aged and older adults are becoming infected with HIV. Clinicians, patients, and society are currently ill-prepared to deal with the biomedical complexities and unique medical and psychosocial challenges associated with the growing aging HIV population.

Aerobic exercise or exercise that speeds up the heart rate lowers CVD risk, and is known to improve physical and mental function with aging, but few well designed studies have reported use of aerobic exercise interventions in PLWH, and no studies have reported whether exercise improves cognitive function in this high risk for CI population. Regular aerobic exercise performed 5 times per week for 150 minutes has also been shown to improve aspects of cognitive function in community-dwelling older adults. Only one exercise study however, has examined the effect of exercise on cognition in PLWH and was limited by a self-reported, unreliable indicator of cognitive status; no studies have reported whether exercise improves cognition in this population using objective assessments, or examined the potential mechanisms involved.

The home-based, 5 day per week moderate intensity walking intervention, the 'Let's Move Program,' has been tested and is effective for lowering CVD risk older caregivers and adults with advanced CVD. The proposed pre-post test pilot study will examine the feasibility of implementing the Lets Move Program among 40 PLWH over 6-months. Participants enrolled in the study will be ≥ 50 years of age, sedentary, have 2 CVD risk factors such as high blood pressure and obesity and demonstrate mild to moderate CI using standardized tests. Motivational Interviewing (MI) will be used to promote exercise confidence and optimize adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 50 and over with 2 CVD risk factors (i.e., obesity, hypertension, hyperlipidemia) who are diagnosed with HIV/AIDS and willing to participate
* English speaking
* live independently and within a 30 mile radius of Atlanta
* not involved in any structured exercise program or exercising 3 or more times per week for a minimum of 30 minutes
* not involved in any weight loss program
* not hospitalized within the last 60-days
* clinically stable (absence of viral load and no active opportunistic infection), on ART 6 months before enrollment and a screening MOCA score ≤ 24 indicating mild cognitive impairment

Exclusion Criteria:

* non sedentary (defined as engaging in > 30 minutes of moderately strenuous exercise 3 times or more a week)
* medical or physical condition that would preclude participation in the exercise component of the study (e.g., severe arthritis or mobility problems, uncontrolled hypertension or diabetes, renal failure, or a history of angina with activity
* ischemic changes or inappropriate BP changes on BL exercise (modified Balke) treadmill test
* on corticosteroids, experiencing acute inflammation at time of baseline or follow-up testing (this will result in rescheduling of testing if no other exclusion criteria apply)
* presence of current opportunistic infection
* any terminal illness
* regular use of anti-inflammatory medications such as non-steroidal anti-inflammatory agents
* women who are pregnant
* severe learning disabilities, intellectual disabilities, psychotic disorders to minimize confounding effects on neurocognitive data
* confounding neuro-medical conditions (e.g., active CNS opportunistic infections, seizure disorders, head injury with loss of consciousness greater than 30 minutes, intracranial neoplasms, stroke with neurological or neuropsychiatric sequelae, and non-HIV-associated dementias)
* active substance abuse and major depression

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-03-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Executive function as measured by stop signal task (SST) of the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 6 months
  SST is a commonly used test of response inhibition. This test consists of two parts. In the first part, the subject is introduced to the press pad, and told to press the left hand button when they see a left-pointing arrow or press the right hand button when they see a right-pointing arrow. There is one block of 16 trials for the subject to practice this. In the second part, the subject is told to continue pressing the buttons on the press pad when they see the arrows, as before, but, if they hear an auditory signal (a beep), they should withhold their response and not press the button.

SECONDARY OUTCOMES:
Executive function as measured by spatial working memory (SWM) of the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 6 months
  SWM is a computerized assessment of working memory and strategy performance. The subject is required to find blue "tokens" in various displayed boxes and use the "tokens" to fill a column on the right side of the screen. Subjects can only find "tokens" in new boxes, therefore they must remember where previous "tokens" were found. SWM scores including number of between errors, number of within errors, and number of double errors range 0-800 and SWM strategy scores range 8-56. Lower scores indicate better performance.
Executive function as measured by attention switching task (AST) of the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 6 months
  AST is a test of the participant's ability to switch attention between the direction or location of an arrow on screen. This test is a sensitive measure of frontal lobe and 'executive' dysfunction. The test begins with an arrow in the centre of the screen which points either to the left or to the right. The participant is introduced to two buttons, one on the left and one on the right, and is asked to press a button corresponding to the direction in which the arrow is pointing.
  After this initial training, the participant is then told that the arrow might appear on the left or the right side of the screen, and depending on the cue given at the top of the screen, the participant must either press the left or right button to indicate on which side of the screen the arrow is displayed, or else press the left or right button to correspond with the direction in which the arrow is pointing.
Memory function as measured by delayed matching to sample (DMS) of the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 6 months
  DMS has 19 outcome measures, assessing latency (the participant's speed of response), the numbers of correct patterns selected, and statistical analysis measuring the probability of an error after a correct or incorrect response.
Memory function as measured by visual recognition memory (VRM) of the Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, 3 months, 6 months
  During VRM, the participant is shown a list of words and then asked to recognize the words they have seen before from a list containing the original words and distractors. The five outcome measures for VRM cover correct and incorrect responses for the recognition and free recall parts of the test.
Information processing speed as measured by choice reaction time (CRT) | Baseline, 3 months, 6 months
  Choice reaction time (CRT) is a computerized assessment that trains the subject in holding down a press-pad and releasing the press-pad in response to stimuli presented on the screen. The task requires the subject to react as soon as a yellow dot appears in one of five locations, and the subject must respond by lifting their hand from the press-pad. This is the reaction time (RT) and ranges from 100 to 5000 msec. Lower scores indicate better performance.
Interleukin 6 (IL-6) Levels | Baseline, 3 months, 6 months
  IL-6 is a pro-inflammatory cytokine known to contribute to the pathogenesis of risk of CVD and CI through inflammation and promotion of endothelial vascular dysfunction. IL-6 is measured by enzyme-linked immunosorbent assay (ELISA) and reported as in picograms per deciliter (pg/dL). Higher concentrations of IL-6 raise CHD risk.
Soluble CD14 (sCD14) Levels | Baseline, 3 months, 6 months
  sCD14 is a marker of monocyte activation, associated with neurocognitive impairment and HIV-associated neurological disorders (HANDs) and higher mortality in PLWH
D-Dimer Levels | Baseline, 3 months, 6 months
  D-Dimer is a marker of procoagulation, associated with increased risk for CVD and neurocognitive decline in older adults. High concentrations of D-dimer have been linked prospectively to onset of CVD and reported as in nanograms per milliliter (ng/mL).
Brain-derived Neurotrophic Factor (BDNF) Levels | Baseline, 3 months, 6 months
  BDNF is a protein that occurs naturally in the hippocampus, cortex, and basal forebrain-areas vital to learning, memory, and higher thinking; an increase in BDNF in animal models and humans is thought to enhance neurogenesis. BDNF is reported as in nanograms per milliliter (ng/mL).
Flow-Mediated Dilation | Baseline, 3 months, 6 months
  Flow-mediated dilation of the brachial artery will be measured using high-resolution ultrasound. Arterial diameter will be measured above the small cavity in the elbow joint from ultrasound images at rest in response to an increase in blood flow to the area.
V02 max | Baseline, 3 months, 6 months
  V02 max is the maximum rate of oxygen consumption as measured during incremental exercise using the Balke treadmill test.
Beck Depression Inventory-II (BDI-II) | Baseline, 3 months, 6 months
  BDI-II is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression. Each answer being scored on a scale value of 0 to 3.
Health-related Quality of Life (HRQoL) | Baseline, 3 months, 6 months
  HRQoL is an assessment of how the individual's well-being may be affected over time by a disease, disability, or disorder.
Exercise Adherence (number of exercise sessions recorded/number of sessions prescribed) × 100) | Baseline, 3 months, 6 months
  Exercise Adherence is the extent to which a patient acts in accordance with the advised interval, exercise dose, and exercise dosing regimen (number of exercise sessions recorded/number of sessions prescribed) × 100.
Steps (measure of walking by a FitBit device) | Baseline, 3 months, 6 months
  Steps is the measure of walking by a FitBit device.
Step Calendar (document participants will be asked to record) | Baseline, 3 months, 6 months
  Step Calendar is a document participants will be asked to record: maximum HR, highest rate of perceived exertion (RPE) during walk, and number of steps walked during the walking sessions.
Borg Rate of Perceived Exertion (RPE) Scale | Baseline, 3 months, 6 months
  RPE is a well-established 15 point (6-20) scale used to measure exertion.
Target heart range (THR) | Baseline, 3 months, 6 months
  THR will be used to monitor the intensity and training response to walking. Target exercise rate will equal peak HR established from CPET (Peak HR) X (0.60 to 0.70). Polar Beat Watch (FT 1) will be used to monitor intensity and duration for the aerobic training.
Exercise Self Efficacy scale | Baseline, 3 months, 6 months
  Exercise Self Efficacy scale is the 18 item scale to measure exercise self-efficacy. Scores range from 0 to 100 with higher scores reflecting greater self-efficacy.
Outcome Expectations for Exercise Scale (OEE) | Baseline, 3 months, 6 months
  OEE is a 9 item scale, with established validity and reliability in older adults and African American's will be used to measure outcome expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gary, RN, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - The Ponce de Leon Center of the Grady Health System, Atlanta, Georgia
  - AbsoluteCARE, Inc., Atlanta, Georgia
  - Emory Hospital Infectious Diseases Clinic, Atlanta, Georgia